CLINICAL TRIAL: NCT01919424
Title: Comparison of the Methacholine PC20 Between the Trudell Aeroeclipse* II Ban Nebulizer and the Wright Nebulizer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Gail Gauvreau, Investigator, McMaster University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HIREB 11-004
Record Dates: First submitted 2013-08-02; First posted 2013-08-09 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Methacholine Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 'The English-Wright nebulizer' (Active Comparator): The English-Wright nebulizer will be used to perform a methacholine challenge.
  Interventions: Drug: Methacholine Chloride; Device: The English-Wright nebulizer
- Trudell AeroEclipse*II BAN nebulizer (Active Comparator): The Trudell AeroEclipse*II BAN nebulizer will be used to perform a methacholine challenge
  Interventions: Drug: Methacholine Chloride; Device: Trudell AeroEclipse*II BAN nebulizer

INTERVENTIONS:
Drug: Methacholine Chloride — Choline ester that acts as a non-selective muscarinic receptor agonist in the parasympathetic nervous system
  Low risk - commonly used to diagnose asthma
Device: Trudell AeroEclipse*II BAN nebulizer — Generates aerosol after a certain inspiratory flow has been reached and then stops nebulization the moment the inspiratory flow falls below this value
  Arms: Trudell AeroEclipse*II BAN nebulizer
Device: The English-Wright nebulizer — Continuous-mode nebuilzer, designed to operate continuously with tidal breathing
  Roxon Medi-Tech, Montreal, PQ, Canada
  Arms: 'The English-Wright nebulizer'

SUMMARY:
This study will compare the methacholine PC20 of two different modern-delivery aerosol systems to determine if one may replace the other for use in clinical settings.

DETAILED DESCRIPTION:
Thirty three asthmatic subjects (>18 years, both sexes) who have stable asthma will be recruited to undergo methacholine challenges for a randomized, crossover, observational study. The objective of this study is to compare the methacholine PC20 of a modern delivery aerosol system, the Trudell AeroEclipse*II BAN nebulizer, to that of the current "gold standard", the English-Wright nebulizer. Subjects will inhale methacholine using both nebulizing systems on separate visits and the PC20 values will be compared. The results from these experiments will give us a better indication of whether the modern AeroEclipse* II BAN nebulizer might be sufficient to replace the current "gold standard" Wright nebulizer in clinical settings.

Baseline Spirometry

Baseline FEV1 and VC will be registered using an electronic spirometer meeting ATS requirements.

Screening

A medical history will be conducted by interview and asthma medications will be reviewed on this V1. Subjects will also undergo a Methacholine Challenge to determine their PC20 and therefore their eligibility into the study.

Methacholine Challenge

Challenges will be carried out after a minimum 8-hour washout of short-acting ß2-agonist. Subjects will perform methacholine challenges on 2 separate days at the same time of day, at least 24-hours apart and all within a 2-week period. At V2, subjects will be randomly assigned to use either the Wright nebulizer or the AeroEclipse*II BAN nebulizer. Methacholine inhalation from the Wright nebulizer will be performed as follows. Subjects are instructed to wear noseclips and to breathe normally from the mouthpiece during the 2-minute inhalation period. Subjects inhale normal saline, then doubling concentrations of methacholine for 2 minutes each always starting at a dose of 0.03 mg/ml. Spirometry is measured with an electronic spirometer meeting ATS requirements. FEV1 is measured at 30 and 90 seconds after each inhalation and the highest FEV1 will be used to calculate the % fall from baseline. There is a 3 minute interval between the end of one inhalation dose and start of the next inhalation dose. The test is terminated when a fall in FEV1 of 20% of the baseline value occurs and the methacholine PC20 is calculated. The same protocol will be applied to methacholine inhalation using the AeroEclipse*II BAN nebulizer with the exception that the 2-minute tidal breathing will be reduced to 20 seconds and the interval between the end of one inhalation dose and start of the next inhalation dose is 3 minutes and 40 seconds. Subjects will return to the lab on V3 to complete a methacholine challenge using the alternate nebulizer from the one used on V2.

DATA ANALYSIS

The methacholine PC20 values will be log-transformed before performing summary statistics. The PC20 values will be compared by paired t-test.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with stable asthma.
* Tidal breathing PC20≤16 mg/mL.
* Baseline FEV1 more than 65% of predicted normal.
* Able to complete 3 methacholine challenges on 3 separate days at the same time of day, at least 24-hours apart and within a 2-week period. (1 during screening and the other 2 during the study)

Exclusion Criteria:

* Airway infection or allergen exposure during the last 4 weeks.
* Exacerbation during the last 4 weeks.
* Change in dosage of inhaled or oral steroids during the last 4 weeks.
* Inhaled salbutamol less than 8 hours prior to testing.
* Inhaled formoterol or salmeterol less than 36 hours prior to testing.
* Antihistamines during the last 48 hours.
* Chronic health conditions that are determined by the principal investigator to be significant (eg cystic fibrosis).
* Smokers
* Pregnant women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2011-04; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Methacholine PC20 of two different aerosol systems | 2 weeks
  To compare the methacholine PC20 of a modern delivery aerosol system, the Trudell AeroEclipse*II BAN nebulizer, to that of the current "gold standard", the English-Wright nebulizer. FEV1 is measured by spirometry following inhalation of increasing concentrations of methacholine. The PC20 is a calculated value of the amount of methacholine required to cause a 20% fall in the subject's FEV1.

CONTACTS AND LOCATIONS:
Overall Officials: Gail Gauvreau, PhD, Principal Investigator — Study investigator
Locations (1):
- McMaster Cardio-Respiratory Research Lab, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] El-Gammal AI, Killian KJ, Scime TX, Beaudin S, Schlatman A, Cockcroft DW, Gauvreau GM. Comparison of the provocative concentration of methacholine causing a 20% fall in FEV1 between the AeroEclipse II breath-actuated nebulizer and the wright nebulizer in adult subjects with asthma. Ann Am Thorac Soc. 2015 Jul;12(7):1039-43. doi: 10.1513/AnnalsATS.201412-571BC. PMID 25871542